CLINICAL TRIAL: NCT02598232
Title: A 24-week, Single-center, Open-label, Clinical Study to Evaluate the Efficacy and Safety of the 1,414nm Nd:YAG Laser System Added to PEN to Further Alleviate Back Pain in a Lumbar Herniated Intervertebral Disc Patient
Brief Title: The Efficacy and Safety of the 1,414 nm Nd:YAG Laser System for Alleviating Back Pain in a Lumbar Disc Patient
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU-DL-14-001
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2016-04

CONDITIONS: Lumbar Herniated Intervertebral Disc
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1,414nm Nd:YAG laser (Experimental): It has high absorption coefficient in water and a short pulse width.
  Interventions: Device: 1,414nm Nd:YAG Laser System

INTERVENTIONS:
Device: 1,414nm Nd:YAG Laser System — It has high absorption coefficient in water and a short pulse width.

SUMMARY:
This study aims to evaluate the efficacy and safety of the 1,414nm Nd:YAG laser system (ACCUPLASTI) added to Percutaneous Epidural Neuroplasty (PEN), a conventional treatment, to alleviate back pain in a lumbar herniated intervertebral disc patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 19-79 years old
* Patients with moderate disability based on the Oswestry Disability Index (ODI), among those diagnosed with a single level of unilateral herniated intervertebral disc among the 3rd-4th and 4th-5th lumbar vertebrae, or the 5th lumbar vertebra-sacral vertebra with back pain or radiating pain in the lower extremities that has been unresponsive to conservative therapy for more than six weeks
* Patients who have language skills enough to answer questionnaires
* Patients who agree to voluntarily participate in this study and to sign the Informed Consent Form, and who are able to participate for the entire period of this study

Exclusion Criteria:

* Patients with a multi-level, far-lateral, or bilateral lumbar herniated intervertebral disc
* Patients who use an electronic medical device for their cardiovascular system
* Patients who have spondylolisthesis in the relevant lesion
* Patients with neurological defects
* Patients who had undergone surgery on the relevant lumbar vertebra
* Patients with cauda equina syndrome
* Patients with congenital spinal deformity
* Patients with spinal fracture
* Patients with spinal infection, tumor, or other form of inflammatory spondylopathy
* Patients with coagulation disorder
* Patients with a history of malignant tumor (except those with a cured tumor and no re- occurrence for the last five years)
* Patients who had participated in another clinical study within 30 days from their screening visit
* Female patients with child-bearing potential who do not agree to use a medically acceptable contraceptive method* for up to 24 weeks after the use of the investigational medical device during this study

  * Medically acceptable contraceptive method: Condom, oral contraceptive pills taken continuously for more than three months, contraceptive injection or implants, intra- uterine contraceptive device, etc.
* Patients who are pregnant or breastfeeding
* Other patients who are considered unfit to participate in this study with clinically significant findings based on the investigator's judgment

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in the Oswestry Disability Index | Day 0, 24 weeks

SECONDARY OUTCOMES:
Change in the Oswestry Disability Index | Day 0, 4 weeks, 12 weeks
Change in the Visual Analogue Scale | Day 0, 4 weeks, 12 weeks, 24 weeks
12-Item Short-form Health Survey | Day 0, 4 weeks, 12 weeks, 24 weeks
Evaluation of the pain level in 4 steps of excellent, good, fair, poor, according to MacNab's Criteria | Day 0, 4 weeks, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Keung-nyun Kim, Professor, Principal Investigator — Severance Hospital

IPD SHARING:
Plan to Share IPD: No